CLINICAL TRIAL: NCT06588088
Title: Cardiorenal, Metabolic and Circadian Effects of Nighttime Eating
Brief Title: Cardiorenal and Metabolic Effects of Nighttime Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koc University Hospital (Other)
Responsible Party: Principal Investigator, Yavuz Erkam Kesgin, Medical Doctor, Resident in Internal Medicine, Koc University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022.093.IRB1.039
Record Dates: First submitted 2024-02-16; First posted 2024-09-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Night Eating Syndrome; Metabolic Syndrome; Cardiorenal Syndrome; Sleep Disorder
Keywords: Night Eating Syndrome; Nutrition; Metabolic Syndrome
MeSH Terms: conditions — Night Eating Syndrome; Metabolic Syndrome; Cardio-Renal Syndrome; Sleep Wake Disorders | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Nutritional study with a single-arm cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early eaters (Placebo Comparator): The diet of these healthy volunteers was such that no calories were consumed after 19.30 in the evening in the first week of the study.
  Interventions: Other: Dietary
- Night time Eaters (Active Comparator): The diet of the same healthy volunteers was 25% of the daily calorie need calculated according to the Harris - Benedict formula was taken, taking into account the night time eating syndrome (NES) criteria, after 20.30 in the evening.
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary — The diet of these healthy volunteers was such that no calories were consumed after 19.30 in the evening in the first week, and in the second week, 25% of the daily calorie need calculated according to the Harris - Benedict formula was taken, taking into account the nighttime eating syndrome (NES) criteria, after 20.30 in the evening.

SUMMARY:
In this study, the investigators are trying to find out of the effect of nighttime eating on metabolism, cardiorenal, hormonal and circadian rhythm, and a study was conducted to examine the effects of diseases that are quite common in internal medicine practice, such as type 2 diabetes mellitus, chronic kidney disease, hypertension, metabolic syndrome and sleep disorders.

DETAILED DESCRIPTION:
The Coronavirus Disease (COVID)-19 pandemic, which emerged in recent years, has deeply affected living conditions and has had an impact on societies on eating habits. As shown by some studies, it has been shown that night sleep habits have changed and night nutrition and calorie intake have increased due to reasons related to staying at home, working remotely, and isolation during the pandemic period. However, some recent studies have shown a relationship between nighttime eating and conditions that predispose to metabolic syndrome, such as obesity and hyperglycemia. At the same time, prospective studies on the details of the cardiorenal and metabolic effects of night feeding behavior, which is one of the important predisposing factors for metabolic syndrome, are quite insufficient. Although the importance of nighttime eating habits has begun to be emphasized in recent years with recent randomized cross-controlled studies on this subject, there are not yet enough prospective studies on this subject. In this respect, studies on nighttime eating behavior, which is common in society, are important.In this study, a cross-over design study was conducted on the effectiveness of nighttime eating on metabolism, cardiorenal, hormonal and circadian rhythm, and a study was conducted to examine the effects of diseases that are quite common in internal medicine practice, such as type 2 diabetes mellitus, chronic kidney disease, hypertension, metabolic syndrome and sleep disorders. The investigators aim to create a new and additional perspective on the management, treatment and follow-up of common diseases and to contribute to raising awareness about night nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being willing to adapt to the desired feeding time and calories
* Body mass index (BMI) is between 18-30
* Not having any systemic disease, not using chronic medication

Exclusion Criteria:

* -<18, >65 years old
* Failure to comply with the regulated nutrition program
* BMI between <18 and >30
* Presence of systemic disease: E.g. Diabetes Mellitus, Chronic Kidney Disease, Coronary Artery Disease, Hypertension etc.
* Inability to have polygraphy
* Chronic drug use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change of the concentration albuminuria in the Nighttime Eating Period | 1 week
  More than 20% increase during night feeding period
Change of the concentration of serum melatonin levels in the Nighttime Eating Period | 1 week
  More than 50% increase during night feeding period
Change of the concentration of serum leptin levels in the Nighttime Eating Period | 1 week
  More than 50% increase during night feeding period
Change of the Concentration of serum ghrelin Levels in the Nighttime Eating Period | 1 week
  More than 50% increase during night feeding period
Change of the concentration of serum total cholesterol, low-density lipoprotein cholesterol, high density lipoprotein cholesterol and triglyceride levels in the Nighttime Eating Period | 1 week
  More than 20% increase during night feeding period
Change of Concentration of serum glucose in the Nighttime Eating Period | 1 week
  More than 10% increase during night feeding period
Change of Concentration of serum insulin in the Nighttime Eating Period | 1 week
  More than 10% increase during night feeding period
Change of concentration of serum Cortisol Level in the Nighttime Eating Period | 1 week
  More than 50% increase during night feeding period
Change of concentration of serum Fibroblast Growth Factor 21 Level in the Nighttime Eating Period | 1 week
  More than 10% increase during night feeding period
Change of the concentration of serum Cytokeratin 18 level in the Nighttime Eating Period | 1 week
  More than 10% increase during night feeding period
Change of value of Apnea Hypopnea Index in the Nighttime Eating Period | 1 week
  The Apnea-Hypopnea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. Apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation to be considered. Combining AHI and oxygen desaturation gives an overall sleep apnea severity score that evaluates both the number of sleep breathing disruptions and the degree of oxygen desaturation (low oxygen level in the blood) during said disruptions.
  The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. The AHI values for adults are categorized as:
  Normal: AHI<5 Mild sleep apnea: 5≤AHI<15 Moderate sleep apnea: 15≤AHI<30 Severe sleep apnea: AHI≥30More than 10% increase during night feeding period

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kanbay, Medical Doctor, Study Director — Koc University, School Of Medicine
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No